CLINICAL TRIAL: NCT05563623
Title: The Beijing Angle Closure Progression Study (BAPS)
Brief Title: The Beijing Angle Closure Progression Study
Status: Recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wu Huijuan, Leader of Glaucoma Group of Ophthalmology Department, Peking University People's Hospital, Peking University People's Hospital
Other Study IDs: PekingUPHOphthalmology001
Record Dates: First submitted 2022-09-26; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Angle-Closure Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- progression group
- non-progression group

SUMMARY:
The Beijing angle closure progression study (BAPS) aims to explore the 5-year incidence of PACS progressing to PAC or PACG and to determine the possible risk factors of disease progression, which may provide the evidence for choosing the accurate strategies in the management of PACS.

DETAILED DESCRIPTION:
Although the global prevalence of primary angle-closure glaucoma (PACG) is less than half that of primary open-angle glaucoma, the risk of serious bilateral visual impairment caused by PACG is three times more than that of primary open-angle glaucoma. PACG is the leading cause of irreversible blindness all over the world, characterized by closure of the anterior chamber angle. Primary angle closure suspect (PACS), the earliest stage of primary angle-closure diseases (PACD), is defined as no less than three quadrants of appositional contact between the peripheral iris and posterior trabecular meshwork on gonioscopy. The progression from PACS to primary angle closure (PAC) was defined as elevated intraocular pressure (IOP) and the presence of peripheral anterior synechiae (PAS). PACG was characterized as PAC together with evidence of glaucomatous optic neuropathy (GON) or glaucomatous visual field defects. It is estimated that by 2040, the number of PACG cases worldwide will reach 32 million, of which Asian cases account for a large proportion. Therefore, a better understanding the natural history of PACD may play an important role in preventing devastating visual impairment.

Previous studies have reported the prevalence of PAC and PACG was 1%-11.3%, but longitudinal reports on its incidence and progression of earlier stages of angle closure that precede PAC/PACG are scarce, especially for Asian population. A Danish study demonstrated that the rate of progression from the condition of shallow anterior chamber to PACG was 16% at ten-year follow-up. Studies in Asia showed that the rate of PACS progress to PAC or PACG was range from 5.3% to 25.5%. And the risk factors of progression included bilateral PACS, smaller angle width, shorter angle open distance, larger iris curvature, and older age. Of note, these studies evaluated the anterior chamber of subjects with examinations including IOLMaster, A scan, and anterior segment-optical coherence tomography (AC-OCT). However, the ultrasound biomicroscopy (UBM), which is most valuable examination in the evaluation of patients with angle closure, was not used. Thus, details such as the volume of the ciliary body, the degree of ciliary anterior rotation, and parameters related to the vitreous zonule (VZ) might have been neglected. In the past, laser peripheral iridotomy (LPI) was considered to be a precaution against progression of PACD, but a few studies postulated that the benefit of prophylactic LPI was limited for PACS. If PACS with high progression risks can be accurately identified, LPI could be applied to high-risk PACS patients rather than all. Therefore, the research on precise risk analysis for PACS progression is imperative.

The Beijing angle closure progression study (BAPS) aims to explore the 5-year incidence of PACS progressing to PAC or PACG and to determine the possible risk factors of disease progression, which may provide the evidence for choosing the accurate strategies in the management of PACS.

ELIGIBILITY:
Inclusion Criteria:

* "Static" gonioscopy identifying 6 or more clock hours of angle circumference in which the posterior (usually pigmented) trabecular meshwork cannot be seen in both eyes with no peripheral anterior synechiae, and normal intraocular pressure (IOP), optic nerve and visual field.
* Able to provide informed consent

Exclusion Criteria:

* Any evidence of primary angle closure (a narrow angle as defined above, but with PAS and/or IOP > 21 mmHg) or primary angle closure glaucoma (visual field defect or glaucomatous optic neuropathy).
* Previous intraocular surgery or laser treatment, such as cataract surgery, laser trabeculoplasty, trabeculectomy, laser peripheral iridectomy, and laser iridoplasty
* Sign of prior acute attack, such as glaucomatous fleck, keratic precipitates, or iris atrophy.
* Anterior segment structural abnormalities shown by examination, such as iris or ciliary body tumor.
* Severe health problems precluding follow-up such as end-stage heart disease, kidney disease, or lung disease, or terminal cancer.
* Severe eye diseases, such as cataract, macular disease, and retinal detachment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary angle-closure suspect who agree to take part in this trial were given a comprehensive baseline examination and who decline will be asked for a reason. Verbal and written informed consent was obtained from every patient. A comprehensive baseline examination will be done for every enrolled subjects. Patients are monitored for 5 years. All examinations that may be related to subjective judgment and manipulation, i.e. Goldmann applanation (GAT), ultrasound biomicroscopy (UBM), gonioscopy, are performed by experienced examiner.
Sampling Method: Probability Sample
Enrollment: 825 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
the progression rate 1 | 6 months
  the rate of acute angle closureanterior synechiae
the progression rate 2 | 6 months
  the proportion of eyes developing peripheral

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beeijing, China

IPD SHARING:
Plan to Share IPD: No